CLINICAL TRIAL: NCT03169062
Title: Evaluation of Coronary Artery Calcification Using Gated Stationary Chest Tomosynthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-1160
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Results first posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- All patients (Experimental): Gated Stationary Chest Tomosynthesis
  Interventions: Device: Gated Stationary Chest Tomosynthesis

INTERVENTIONS:
Device: Gated Stationary Chest Tomosynthesis — The technologist will comfortably position the patient laying face up on the imaging table. EKG leads will be placed in appropriate positions to derive an EKG signal. The EKG will be used to trigger the image collection. The subject will be asked to hold his or her breath for 25-30 seconds during the scan. Total patient preparation and imaging time should not exceed 20 minutes.

SUMMARY:
The purpose of this study is to propose a new method for evaluating coronary artery calcium scores (CACS) in individuals with coronary artery disease.

DETAILED DESCRIPTION:
The proposed research, if successfully implemented, will result in a new method for evaluating coronary artery calcium scores (CACS) in individuals with coronary artery disease. Using the Cardiac Gated Stationary Chest Tomosynthesis (CG-SDCT) system the imaging dose for a a full tomosynthesis scan is expected to be only 10% of that from a low-dose CT. The targeted imaging time of 25-30 seconds is 1/2 of that from a current commercial DCT system at the same imaging dose. As with current commercial DCT systems, our s-DCT system will expose patients to less radiation and deliver comparable data for CACS. CG-SDCT will likely result in accurate CAC scoring and allow for a more complete patient risk assessment as compared to Framingham risk scoring alone.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: ≥18 years of age
2. Intermediate Framingham Risk Score of 10 to 20% risk over the next 10 years
3. Previous non-contrast enhanced chest CT in a time frame that will accommodate experimental imaging (CG-SDCT) within 4 weeks. This imaging may have already been completed at the time of enrollment or may be scheduled in the future at the time of enrollment.
4. IRB written informed consent obtained and signed Exclusion Criteria
5. Negative urine pregnancy test in women of child-bearing potential (WCBP) within 1 week prior to s-DCT.

Exclusion Criteria:

1. Unable to provide consent
2. Pregnant or lactating
3. BMI > 33 (Patient who may not fit on a 35 x 35 detector) (Images are not clear on subjects who have a greater than 33 BMI)
4. Previous history of MI or thoracic surgery.
5. Disability that could interfere with the scanning process, non-ambulatory or unable to hold their breath for up to 30 seconds.
6. Planned procedures or therapies in between non-contrast CT scan and study Chest tomosynthesis scan, e.g., line placement in the chest region, biopsy, etc.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yueh Lee, M.D, Principal Investigator — University of North Carolina of Chapel hill
Locations (1):
- University of North Carolina of Chapel hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Patients
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 76 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Comparison of CT Derived CACS and Tomosynthesis Scores Correlation
Description: Linear regression and Bland-Altman analysis will be used to examine the relationship between the CT derived CACS and tomosynthesis scores to determine the correlation
Time Frame: 1 year
Population: Visualization of coronary artery calcium was limited given the small effective angular span of the current hardware, thus calcium scoring was not performed. Since calcium scoring could not be performed, the planned analysis could not be conducted.
Arm/Group | All Patients
Number analyzed (Participants) | 0

2. Secondary Outcome: Mean Correlation Coefficient of Gating
Description: The 30 ms cardiac EKG trace will be extracted for each of the projections. Then, a Pearson correlation coefficient will be calculated for each of the projections relative to the first x-ray projection. The mean of the Pearson correlation coefficients will then calculated and served as an estimate of the timing precision of each projection set for each patient. The mean and standard deviation of the correlation coefficients will be reported.
Time Frame: At the conclusion of all data collection, 6 months post study completion
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | All Patients
Number analyzed (Participants) | 10
unitless | 0.87 (0.09)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT03169062/Prot_SAP_000.pdf